CLINICAL TRIAL: NCT06083818
Title: Therapeutic Exercise Protocol for the Prevention of Anterior Cruciate Ligament Injuries in Female Football Players With Dynamic Knee Valgus
Brief Title: Anterior Cruciate Ligament Injury Prevention Protocol in Female Football Players With Dynamic Knee Valgus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Amanda Coves García (Other)
Responsible Party: Sponsor-Investigator, Amanda Coves García, Principal Investigator, Universidad Miguel Hernandez de Elche
Organization: Universidad Miguel Hernandez de Elche (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 04122022
Record Dates: First submitted 2023-07-25; First posted 2023-10-16 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: Knee Injuries; Female; Football
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Knee Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blind masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants in this group will undergo a conventional physical preparation programme.
  Interventions: Other: Placebo - Conventional fitness programme
- ACL injury prevention protocol (Experimental): Participants in this group will undergo a specific 12-week prevention protocol.
  Interventions: Other: Application of an anterior cruciate ligament injury prevention protocol for female football players with dynamic knee valgus for 12 weeks.

INTERVENTIONS:
Other: Application of an anterior cruciate ligament injury prevention protocol for female football players with dynamic knee valgus for 12 weeks. — 12-week ACL Injury Prevention Protocol
  Arms: ACL injury prevention protocol
Other: Placebo - Conventional fitness programme — Conventional training and physical preparation programme
  Arms: Placebo

SUMMARY:
Introduction: Women's football has experienced exponential growth over the last ten years. Its popularity is associated with an increase in anterior cruciate ligament injuries (ACL). They constitute a major current problem as they account for 43% of the injury burden during the sport season. Despite existing training programmes, no uniform criteria have been established to design a precise intervention protocol, with specific tasks linked to women's football, nor has it been proposed to optimise current programmes.

Objective: To evaluate the efficacy of a comprehensive and specific training protocol focused on female football players with dynamic knee valgus (DKV) to prevent ACL injuries.

Methodology: Randomised, double-blind, single-centre clinical trial protocol scheduled for the 2023-2024 season of women's football. There will be 2 groups: a group that will follow a specific ACL injury prevention protocol and a control group. The intervention period will last 12 weeks. Measurements will be taken at 3 time points. The biomechanics of the lower extremities, the dynamics of jumping and landing, as well as the pre and post training satisfaction of the players will be evaluated. Image capture and processing systems will be used in addition to tests such as the drop vertical jump test (DVJ), the LESS scoring system, among others.

Future expectations: This protocol aims to be one of the first to implement an ACL injury prevention programme for women football players with DKV. Despite the scarcity of research in this area, studies support beneficial effects at a preventive level.

ELIGIBILITY:
Inclusion Criteria:

* Female football players registered and federated in the corresponding team.
* With an age range between 18 and 35 years old.
* Minimum experience of one year playing football.
* With DKV presence.

Exclusion Criteria:

* Subjects with previous ACL or other ligamentous injury to the knee.
* Subjects with a history of lower extremity injury resulting in surgery during the six months prior to the study.
* Players with chronic illnesses that may affect test results.
* Subjects who played other sports at a professional level.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
CHANGING RISK FACTORS | 12 weeks
  modification of risk factors such as dynamic knee valgus
MOTOR CONTROL | 12 weeks
  Changes in motor control not only of the lower limbs, but also of the lumbo-pelvic complex using software and imaging systems that measure joint alignments.
SPORT PERFORMANCE | 12 weeks
  Tactical and technical changes are expected on the pitch as well as improvements in the sporting performance of the players through dynamic evaluations with imaging and video systems as well as speed and agility tests by monitoring joint stability.
KNEE JOINT BIOMECHANICS | 12 weeks
  Changes in neuromuscular control of the knee using imaging and force plate assessments to monitor lower limb alignment and areas of increased reaction force.
SPORTSWOMEN SATISFACTION | 12 weeks
  Changes in the incidence of injuries among female football players using the SF-12 satisfaction scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Miguel Hernandez University, Sant Joan d'Alacant, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data concerning the age, height and weight of the participants will be shared, as well as the variables that will be measured for the subsequent execution of the study.
  A statistical analysis of the required variables will be carried out, in addition to explaining the data analysis system using statistical programmes. Informed consent will also be obtained from each of the participants in the study, specifying the collection of personal data for research and teaching purposes.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Since the completion of the study and reporting of the study by publishing it in an international journal
Access Criteria: Anyone who subscribes to the journal and who has access to the articles published in the journal

REFERENCES:
- [Background] Coves-García A, Lozano-Quijada C, Poveda-Pagán EJ. Strategies for the prevention of anterior cruciate ligament injuries in female athletes with dynamic knee valgus. Systematic review. Physiotherapy. doi:https://doi.org/10.1016/j.ft.2023.04.002.
- [Derived] Garcia AC, Pagan EJP. Therapeutic exercise protocol for the prevention of anterior cruciate ligament injuries in female soccer players with dynamic knee valgus (RCT). Trials. 2025 Jan 29;26(1):29. doi: 10.1186/s13063-025-08736-7. PMID 39881313

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT06083818/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT06083818/ICF_001.pdf